CLINICAL TRIAL: NCT06067243
Title: Valutazione Della Performance Diagnostica di MRI 3T Con Tecnica T2 Mapping e Correlazione Intraoperatoria Artroscopica Nella Patologia Condro-labrale Dell'Anca: Studio Interventistico di Validazione di Tecniche Diagnostiche (HPI MRI 3T)
Brief Title: Diagnostic Performance of 3T MRI T2 Mapping Technique in Chondro-labral Pathology of the Hip, Correlated With Intraoperative Arthroscopic Findings: Interventional Diagnostic Technique Validation Study (HPI MRI 3T)
Status: Withdrawn | Type: Observational
Why Stopped: No patients
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: CE-AVEC 577/2020/Sper/IOR
Record Dates: First submitted 2023-09-05; First posted 2023-10-04 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Hip Injuries and Disorders; Hip Arthrosis
Keywords: 3T MRI; labral and chondral lesions; hip arthroscopy
MeSH Terms: conditions — Hip Injuries; Disease; Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIP MRI-3 T: Young patients with coxalgia and clinical and imaging suspect for cartilage and/or labral lesion of the hip
  Interventions: Diagnostic Test: T2 mapping 3T MRI + hip arthroscopy

INTERVENTIONS:
Diagnostic Test: T2 mapping 3T MRI + hip arthroscopy — 1. 3T MRI
  2. hip arthroscopy

SUMMARY:
The goal of this observational study is to evaluate the diagnostic performance of the T2 mapping technique of the following 4 MRI scans in detecting hip chondro-labral lesions in comparison with intraoperative arthroscopic findings: 1) basal 3T MRI with T2 mapping technique, 2) 3T MRI with T2 mapping technique and limb traction; 3) 3T arthro-MRI with T2 mapping technique; 4) 3T arthro-MRI with T2 mapping technique and limb traction.

DETAILED DESCRIPTION:
This study will evaluate the role of T2 mapping technique in the diagnosis of chondral and labral lesions of the hip. In particular, the following 4 types of MRI scan will be compared to each other and with intraoperative arthroscopic findings:

* Basal 3T MRI without contrast
* 3T MRI with limb traction
* Arthro-RM 3T after intrarticular gadolinium and local anesthetic injection under ultrasound control
* Arthro-RM 3T after intrarticular gadolinium and local anesthetic injection under ultrasound control + limb traction.

The primary endpoint is to:

* assess the diagnostic performance of baseline 3T MRI with T2 mapping technique in terms of sensitivity, specificity, PPV, and NPV in the diagnosis of hip labral lesions, according to Philippon's classification, and chondral lesions according to modified Outerbridge classification,
* compare the diagnostic performance between all the mentioned above scans.

The secondary endpoint is to evaluate the sensitivity, specificity, PPV and NPV of 3T MRI with longitudinal traction of the lower limb in detecting, localizing and grading chondral lesions of the coxo-femoral joint.

The present study will involve 30 young patients with coxalgia non responding to conservative treatment and referable to a chondro-labrum injury based on clinical and imaging examinations.

Patients will undergo RM diagnostic protocol and will receive hip arthroscopy within the next 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic localized chondro-labral lesion requiring arthroscopic treatment
* Consent to conduct the study
* BMI<30

Exclusion Criteria:

* Patients unable to read or understand the patient information and consent forms;
* Previous surgery on the same hip;
* Coxarthrosis ≥ 2 according to Tonnis;
* Acetabulum and/or proximal femur fractures;
* Presence of psychological disorders, which might interfere with their ability to undergo the 4 MRI examinations;
* Known sensitivity to gadolinium;
* BMI ≥ 30;
* Current infections;
* Tumors;
* Metabolic disorders;
* Presence of peripheral neurological disorders such as pudendal neuralgia, peroneal neuralgia, neuralgia sciatica that traction may risk worsening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young with symptomatic localized chondro-labral lesion requiring arthroscopic treatment
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
T2 mapping 3T MRI | At baseline (Day 0)
  * Grade of cartilage lesions according to modified Outerbridge classification;
  * Grade of labrum lesions according to Philippon's classification;
  * Localization of cartilage lesions according to the clock system;
  * Localization of labrum lesions by the ROI (Region Of Interest) method.
Hip arthroscopy | Within 6 months from day 0
  * Grade of cartilage lesions according to modified Outerbridge classification;
  * Grade of labrum lesions according to Philippon's classification;
  * Localization of cartilage lesions according to the clock system;
  * Localization of labrum lesions by the ROI (Region Of Interest) method.
Data comparison | Within 21 months from beginning of the study
  In the postoperative phase, the intraoperative findings will be compared with the preoperative findings of the 4 MRI types by proceeding to calculate their sensitivity, specificity, PPV, NPV in relation to the degree and location of chondro-labral lesions of the hip.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No